CLINICAL TRIAL: NCT06046300
Title: Investigation of the Relationship Between Trunk Position Sense and Muscle Activation, Balance and Quality of Life in Individuals With Transtibial Amputation
Brief Title: The Relationship Between Trunk Position Sense and Muscle Activation, Balance and Quality of Life in Amputees
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Semra Topuz, PT, MSC, Clinical Professor, Hacettepe University
Other Study IDs: GO 21/1104
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Amputation; Muscle Activation; Balance; Quality of Life; Sense of Control
Keywords: Transtibial amputation; Sense of position; Muscle activation; Balance; Quality of Life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amputees: Individuals with a transtibial amputation
  Interventions: Diagnostic Test: Investigation of the relationship between trunk position sense and muscle activation, balance and quality of life in individuals with transtibial amputation.
- Healthy: Healthy individuals
  Interventions: Diagnostic Test: Investigation of the relationship between trunk position sense and muscle activation, balance and quality of life in individuals with transtibial amputation.

INTERVENTIONS:
Diagnostic Test: Investigation of the relationship between trunk position sense and muscle activation, balance and quality of life in individuals with transtibial amputation. — It is aimed to investigate whether the trunk position sense, including the trunk right and left sides of the individuals with transtibial amputation, is affected and the relationship between trunk position sense and muscle activation, balance and quality of life.

SUMMARY:
This study was planned to examine the relationship between trunk position sense and muscle activation, balance and quality of life in individuals with transtibial amputation. Individuals with unilateral transtibial amputation who have been using prostheses for at least 1 year and volunteered to participate in the study, as well as healthy individuals with similar demographic characteristics will be included in the study. The number of cases considered to be included in the study will be obtained from the statistical analysis of the results of the pilot study to be conducted with 5 individuals, since there is no study on the subject. The power of the study will be determined as 0.80. After determining the number of individuals to be included in the study group, a control group will be formed with the same number of healthy individuals. The study will be terminated when the determined total number of participants is reached. Body position sense, trunk muscle activation, static and dynamic balance performances and quality of life of all individuals will be evaluated. Body position sense of individuals with "Dualer IQ Pro Digital Inclinometer" device, trunk muscle activation with "Delsys Trigno IM wireless surface electromyography (sEMG) system", balance with "Bertec balance platform", balance and functional mobility with "Berg Balance Scale (BDI) ", "Timed Up and Go Test (SKYT)" and "Modified Star Excursion Test (SEBT)" and quality of life will be evaluated with "Trinity Amputation and Prosthesis Experience Scale (TAPES)". As a result of our study, investigators think that it will contribute to the current scientific knowledge about the somatosensory and biomechanical mechanisms underlying the abnormalities that occur in the trunk after transtibial amputation, to determine whether the trunk position sense of individuals with transtibial amputation is affected or not, and to determine the relationship between trunk position sense and muscle activation, balance and quality of life.

DETAILED DESCRIPTION:
Amputation is a major trauma that significantly disrupts the biomechanics of the musculoskeletal system, results in serious physical and psychological losses, and affects the quality of life, social and professional life of the individual.

Following lower extremity amputation, somatosensory input, muscle activity, and joint mobility decrease in the amputated part of the extremity.

The ability to maintain postural stability is one of the most important aspects of our daily lives.

While standing, the postural control system adjusts the center of pressure and gathers inputs from the visual, vestibular, and somatosensory systems (i.e. proprioceptive and cutaneous senses) to maintain the center of gravity on the base of support.

The ability to maintain balance is severely impaired following lower extremity amputation.

As the stump fails to compensate for the lack of foot and ankle as a proprioceptive organ, the postural control system is reprogrammed and compensatory mechanisms are developed to prevent weight-bearing asymmetries, somatosensory loss, reduced support surface, and increased joint stiffness.

These changes are also reflected in changes in neuromuscular motor output, such as postural sway during standing.

Although used prostheses are an alternative to partially reduce deficiencies, current prosthetic technologies do not provide enough sensory feedback.

Persons with lower extremity amputations exhibit abnormal trunk movement during functional tasks than non-injured persons.

As shown in studies, an asymmetrical posture and balance problem occurs in individuals with amputation.

The resulting asymmetry can be associated with chronic neuromuscular problems such as back and extremity pain, vascular diseases, and early arthritis.

Controlled trunk movement is essential for balance and stability while walking. Individuals with lower extremity amputations often exhibit abnormal trunk movement, but the underlying mechanisms are not well understood.

Lower extremity amputation results in loss of muscles, tendons, ligaments and joint capsule, severely affecting the lower extremity and thus body function.

These structures are not only essential for movement, they also function as sensory receptors, and when lost, proprioception suffers.

It includes conscious proprioception, kinesthesia, strength sense, and joint position sense.

Several studies have investigated changes in proprioception in individuals with transtibial amputation and have presented different results.

Fontes et al. concluded that asymmetric body weight distribution was not accompanied by a decrease in knee proprioception in transtibial amputees.

Latanioti et al. They stated that when joint position sense at 15° was evaluated, stump proprioceptive knowledge was not significantly affected after knee amputation and prosthesis application, and the loss of knee sensory receptors in these individuals was compensated by alternative mechanisms.

Liao and Skinner concluded that there is a significant difference in knee joint proprioception between prosthetic and intact limbs in persons with below-knee amputation.

Eakin et al. They designed a proprioception measurement system to evaluate lower extremity knee joint proprioception in 10 above-knee amputees.

The system allowed subjects to be tested in a position simulating the late swing phase of gait.

The ability to repeat the lower extremity positions specified for the intact and prosthetic extremities of the subjects was recorded for the detection of slow passive movement.

As a result of the study, a significant difference was detected between the passive motion detection threshold of the amputated and intact extremities; however, they stated that there was no significant difference between passive motion reposition of amputated and intact extremities.

This finding demonstrates the importance of hip joint motion appreciation when these motions are relevant in the proprioception of the prosthetic knee joint of amputees.

However, prosthetic limb passive motion positioning error decreases with age, which may improve amputees' ability to use the remaining lower extremity proprioceptive mechanisms to compensate for the loss of anatomical knee joint structures.

There are many studies in the literature examining position sense, muscle activity, balance and quality of life in individuals with transtibial amputation.

However, studies have focused on the lower extremities. Individuals with transtibial amputation often have abnormal trunk movement, but the mechanisms underlying this abnormality in terms of trunk are not well understood.

Information on trunk muscle activity and trunk position sense in individuals with transtibial amputation is very limited.

In the current literature, the trunk position sense of individuals with transtibial amputation and the relationship of trunk position sense with muscle activation, balance and quality of life.

Therefore, in this study, it is aimed to investigate whether the trunk position sense, including the trunk right and left sides of the individuals with transtibial amputation, is affected and the relationship between trunk position sense and muscle activation, balance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

For Transtibial Amputation Group;

* Having a traumatic unilateral transtibial amputation,
* Using prosthesis for at least 1 year,
* K2 and K3 functional classification according to K level,
* Between the ages of 18-45,
* Having received standard physiotherapy methods (prosthesis training),
* It was determined as individuals who volunteered to participate in the study. For the Healthy Group;
* Between the ages of 18-45,
* Having similar demographic characteristics with the individuals in the transtibial amputee group,
* No neurological and/or orthopedic problems,
* Individuals who agreed to participate in the study voluntarily.

Exclusion Criteria:

For both groups;

* Having hip, knee or ankle joint limitation,
* Having muscle shortness that prevents walking and other activities,
* Having a history of falling in the last 1 year,
* Body mass index (BMI) >30 kg/m²,
* Individuals using a walking aid. For the Amputation Group;
* Having phantom pain,
* Individuals with any disease or systemic health problem that may affect their gait other than amputation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study group consisted of individuals with transtibial amputation who volunteered to participate in the study and came to Hacettepe University Faculty of Physical Therapy and Rehabilitation, Prosthesis-Orthotics and Biomechanics Unit and Bilim Orthotics Prosthesis Center; The control group will consist of healthy individuals in the immediate vicinity who volunteered to participate in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Trunk Position Sense measurement | 30 minutes
  Thanks to dual-sensor measurement with Dualer IQ Pro Digital Inclinometer, spine evaluations can be made by collecting easy and reliable data. The device is recommended by the American Medical Association (AMA). It is a calibrated device with a 1 degree margin of error, used in the measurement of joint range of motion and position sense in the clinic. It determines the potential difference between the two end heads and converts this potential difference to the corresponding joint angle to measure the range of motion of the spine and limbs without a computer.

SECONDARY OUTCOMES:
Trunk Muscle Activation measurement | 30 minutes
  Evaluation of erector spinals (m. Longissimus, m. iliocostalis), lumbal multifidus, rectus abdominis and external oblique muscle activations will be performed using the Delsys Trigno IM (Delsys Inc. Natick, Massachusetts, USA) wireless surface electromyography (sEMG) system. The evaluation of trunk muscle activation will be made with the Bertec balance platform during the balance evaluation, and the surface electrodes that will be used to record the electromyography (EMG) signals of the trunk muscles will be selected and applied in accordance with the recommendations of SENIAM (Surface ElectromyoGraphy for the Non-Invasive Assessment of Muscles).

OTHER OUTCOMES:
Balance measurement | 30 minutes
  While the balance assessments of the cases are made using the Bertec BalanceCheck Screener™ BP5050 20x20 inc platform (Bertec BP5050 balance plate platform; Bertec, Corp., Columbus, OH, USA), muscle activations will be evaluated with superficial EMG at the same time as the assessment. The Bertec balance platform is a three-component platform that aims to objectively measure instantaneous changes in the vertical force and center of pressure (Center of Pressure-CoP).
Quality of Life measurement | 30 minutes
  The Turkish version of the Trinity Amputation and Prosthesis Experience Scale (TAPES), a versatile assessment tool developed to determine prosthesis satisfaction and compliance level in amputees, will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Ulger, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No